CLINICAL TRIAL: NCT03318276
Title: A Multicenter, Randomized, Double-Blind, Active-Controlled, Parallel Group and Phase III Clinical Trial to Evaluate in Efficacy and Safety of SID142 in Patients With Chronic Artery Occlusive Disease
Brief Title: Clinical Trial to Evaluate Efficacy and Safety of SID142 in Patients With Chronic Artery Occlusive Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SID142_ATP_III_2015
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2018-09

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SID142 (Experimental): Patients administrate SID142 (Cilostazol 200mg, Ginkgo biloba leaf extract 160mg) once a day for 12 weeks
  Interventions: Drug: SID142
- Rinexin® Tab (Active Comparator): Patients administrate Rinexin® Tab (Cilostazol 100mg, Ginkgo biloba leaf extract 80mg) twice a day for 12 weeks
  Interventions: Drug: Rinexin® Tab

INTERVENTIONS:
Drug: SID142 — SID142 is administrated to patients with PAD for 12 weeks
  Other Names: Placebo (For Rinexin® Tab)
  Arms: SID142
Drug: Rinexin® Tab — Rinexin® Tab is administrated to patients with PAD for 12 weeks
  Other Names: Placebo (For SID142)
  Arms: Rinexin® Tab

SUMMARY:
Rinexin® Tab (Cilostazol 100mg, Ginkgo biloba leaf extract 80mg) has been widely used as an anti-platelet agent for the treatment of PAD. SID142 is a new controlled-release product improved patient's convenience and disadvantage of dosage regimen of previous drug. The aim of this study was to compare the efficacy and safety of SID142 and Rinexin® Tab in patients with PAD

DETAILED DESCRIPTION:
This clinical trial is 12 weeks, multicenter, randomized, double-blind, parallel group, phase 3 study which registered patients in total 19 institutions appointed as national clinical trial institution, it was conducted by receiving IRB(institutional review board) approval from each institutions.

Target patients were aged over 20 years old male or female lower limb peripheral artery occlusion patients with fontaine stage II/III, who has lower limb pain. Lower limb pain degree is over 40 mm evaluated by VAS at screening, and ABI (ankle-brachial index) ≤0.9 or stenosis rate over >50%, diagnosed with PAD and voluntarily agreed to participate in clinical study and signed study consent form. Study subjects who met subjects criteria and recruited were total 170 subjects. Selected subjects were stratified by 1:1 ratio and randomly assigned to investigational product or comparator.

Investigational product was SID142 and comparator was Rinexin® Tab (Cilostazol 100mg, Ginkgo biloba leaf extract 80mg). Administration period to subjects was 12 weeks, study group took investigational product, SID1421 tab once(morning) and took placebo 1 tab/once, 2 times/day, and comparator group took investigational product, Rinexin® Tab 1 tab/once, 2 times/day and took placebo 1 tab once(morning).

Efficacy and Safety Assessment Parameter Subjects visited at 4, 8, and 12 weeks including baseline visit (visit 2) at 4 weeks interval and took efficacy and safety.

Variation in lower limb pain (VAS) comparing baseline with 12 weeks point as a primary efficacy Assessment parameter, variation in lower limb pain (VAS) comparing baseline with 4, 8 weeks, ankle brachial pressure index (ABI), ankle systolic pressure (ASP), Maximum Walking Distance (MWD), Pain Free Walking Distance (PFWD), andInvestigator's global assessment (5-point scale) as secondary efficacy assessment parameters, efficacy was measured. Pain and coldness test was measured using pain and coldness felt by subject 24 hours prior to the visit, MWD and PFWD was measured only on subjects who was determined to be possible to measure. Also, adverse event, laboratory test, vital sign, were conducted for safety assessment. Physical test and vital sign were conducted at screening visit, administration begins, 4, 8, and 12 weeks and urine pregnancy test and laboratory test were conducted at screening visits and 12 weeks. ECG test was conducted at screening visit, 4, 8, and 12 weeks after. Laboratory test criteria were hematological test, blood chemical test, blood coagulation test and urine test.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female outpatients over 20years of age
2. patients confirmed to have PAD

   * ABI ≤0.9
   * Occlusion rate>50%
3. LE PAD with Fontaine stage II/III
4. LE pain VAS≥40mm at screening

Exclusion Criteria:

1. Patients who underwent vascular surgery or endovascular procedure for PAD within 1month prior to study. Patients who need vascular surgery or endovascular procedure for PAD during this study also should be excluded.
2. Patients with peripheral neuropathy.
3. Patients with ischemic heart diseases or underwent percutaneous transluminal coronary angioplasty or coronary artery bypass graft within 6 months prior to study.
4. Patients who has diagnosed cerebrovascular diseases within 6 months prior to study.
5. Patients with hemorrhage or predisposition to hemorrhage at screening visit.
6. Uncontrolled hypertension defined as ≥ 180 mmHg of systolic blood pressure or ≥ 110 mmHg of diastolic blood pressure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Variation in lower limb pain (VAS) | 12 weeks
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure lower limb pain that is believed to range across a continuum of values. The amount of pain that a subject feels ranges across a continuum from none to an extreme amount of pain.
  VAS is a 100mm horizontal line. The patient marks on the line the point that they feel represents their perception of their state.
  The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the subject marks. The higher the score, the more severe the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Donghoon Choi, Principal Investigator — Yonsei University College of Medicine, Severance Cardiovascular Hospital
Locations (1):
- Yonsei University College of Medicine, Severance Cardiovascular Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kook H, Yu CW, Choi D, Ahn TH, Chang K, Cho JM, Kim SJ, Park CG, Cho DK, Kim SH, Lee HC, Jin HY, Chae IH, Kwon K, Ahn SG, Kim JH, Lee SR, Kim JS, Kim SY, Lim SW. Efficacy and Safety of SID142 in Patients With Peripheral Arterial Disease: A Multicenter, Randomized, Double-Blind, Active-Controlled, Parallel-Group, Phase III Clinical Trial. Clin Ther. 2022 Apr;44(4):508-528. doi: 10.1016/j.clinthera.2022.01.016. Epub 2022 Apr 9. PMID 35410753